CLINICAL TRIAL: NCT05950685
Title: Development of a Screening Tool for Prediction of Long-term Arm Morbidity Following Breast Cancer Surgeries and Treatments
Brief Title: Prediction of Long-term Arm Morbidity Following Breast Cancer Surgeries and Treatments
Status: Completed | Type: Observational
Sponsor: Ifat Klein (Other)
Collaborators: Ben-Gurion University of the Negev (Other)
Responsible Party: Sponsor-Investigator, Ifat Klein, Physical therapy coordinator of the field of breast cancer patients treatments, Assuta Medical Center
Organization: Assuta Medical Center (Other)
Other Study IDs: 0019-22ASMC
Record Dates: First submitted 2023-03-19; First posted 2023-07-18 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2024-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Background: Breast cancer (BC) treatments usually include a combination of surgery, chemotherapy and radiation. These life-saving treatments cause high percentages of arm morbidity, which often lasts for months, or develops months after surgery. Arm and shoulder morbidity includes prolonged pain, restriction of movement, limitation of function and lymphedema (chronic progressive edema). All of these morbidities affect the quality of life (QOL) of the recovering patients and require lengthy care. Early detection of patients at risk and provision of proactive treatment can improve the recovery process from surgery and oncology treatments.

Aim: To develop a screening tool for the early identification of women at high risk for prolonged arm morbidity following BC treatments (persistent pain, lymphedema, function deficits and decreased range of motion), validate the tool, and examine the efficiency of intervention based on the the use of the tool.

DETAILED DESCRIPTION:
The development and the assessment of the screening tool will conduct in three stages:

1. Systematic review and meta-analysis to identify from the literature risk factors for lymphedema, prolong pain, decreased range of motion (ROM), quality of life (QOL) and function after breast cancer (BC) treatments and surgery. Intended to understand which factor could be included in the screening tool.
2. Development of the screening tool (study no. 1)- cross section study that will examine which of the risk factors found in the literature review/ meta-analysis will enter the tool. Women up to 3 years after BC surgery will be evaluated for arm morbidity (pain, lymphedema, limitation of movement and limitation of function), and their association to the risk factors, using an online questionnaire.
3. A small cohort study (study no. 2)- Aimed to validate the screening tool. The study will be conducted at the hospital's oncology institute, and will recruit BC survivors who come for routine follow-up six months till three years after surgery. Patients will be asked to answer an online questionnaire, in addition, limb volume tests, strength and ROM will be performed at the clinic. A comparison will be made between the physical parameters that indicate the morbidity of the arm and the score found in the screening tool.
4. A small prospective study (study no. 3)- The main goal of this study is to examine whether the use of the new questionnaire by the patients themselves will; A) affect the percentage of arrival to physical therapy (PT) treatments, B) will affect morbidity rates.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-75
* Independent
* Speaking Hebrew and Russian

Exclusion Criteria:

* Patients who reported that from the time elapsed from the surgery they underwent additional surgery or an injury affecting the function/ pain of the arm.
* Patients suffering from advanced metastatic disease, or background diseases that limit function.
* Lymphedema prior to surgery.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — breast cancer patients
Study Population: Breast cancer patient six months till three years after surgery
Sampling Method: Non-Probability Sample
Enrollment: 1602 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
QuickDASH questionnaire | 18 months
  a shortened version of the The Disabilities of the Arm, Shoulder and Hand (DASH), that contains 11 items measuring an individual's ability to complete tasks, absorb forces, and severity of symptoms. The QuickDASH tool uses a 5-point Likert scale from which the patient can select an appropriate number corresponding to her severity/function level. The the scores range from 0 (no disability) to 100 (most severe disability).
Numeric pain rating scale | 18 months
  Pain scale reported by patients with rage of 0(no pain)-10(the worst possible pain imaginable).
The Godin-Shephard Leisure-Time Physical Activity | 18 months
  divides the effort levels into light/ mild, moderate, strenuous and multiply by time per week.

SECONDARY OUTCOMES:
Number of patients diagnosed with lymphedema | 18 months
  Diagnosis of lymphedema by a doctor / physical therapist
Shoulder range of motion | 18 months
  Using DR Goniometer App evaluating ranges of motion in degrees between 0 (no range) to 180 (full range)

CONTACTS AND LOCATIONS:
Overall Officials: Merav Ben- David, Professor, Principal Investigator — Assuta Medical Center
Locations (1):
- Assuta medical center, Tel Aviv, Israel, Israel